CLINICAL TRIAL: NCT06198270
Title: Effects of Neuromuscular Training With K-tape on Pain, Range of Motion and Balance in Footballer With Ankle Sprain
Brief Title: Effects of Neuromuscular Training With K-tape in Footballer With Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/33
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Ankle Sprains; Proprioception; Pain; Balanced
Keywords: ankle sprain; neuromuscular training; closed kinetic chain; Balance; Functions
MeSH Terms: conditions — Ankle Injuries; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close Kinetic Chain Exercise (Other): Control Group (Close Kinetic Chain Exercise)
  Interventions: Other: Closed Kinetic Chain Exercise
- Neuromuscular training with K-Tape (Experimental): Experimental Group (Neuromuscular training with K-Tape
  Interventions: Other: Neuromuscular Training with K Tape

INTERVENTIONS:
Other: Closed Kinetic Chain Exercise — Closed chain exercise plan of 5 exercises, 10reps x 3sets of each, 3 days in a week for 4-weeks, all values measured before and after 4-weeks.
  Arms: Close Kinetic Chain Exercise
Other: Neuromuscular Training with K Tape — Neuromuscular training plan of 5 exercises, 10reps x 3sets of each, 3 days in a week, for 4-weeks, all values measured before and after 4-weeks. Just After the session k-tape applied.
  Arms: Neuromuscular training with K-Tape

SUMMARY:
This randomized controlled trial, conducted at the Pakistan Sports Board in Lahore from March to August 2023, investigates the impact of neuromuscular training with K-Tape on pain, range of motion, and balance in footballers with grade I and II ankle sprains. A total of 30 male participants aged 18-30, engaged in sports for at least one year with weekly training durations of 15-20 hours, are included in the study through a non-probability convenient sampling technique. The participants are divided into two groups: Group A (Control) receiving closed-chain exercises and Group B (Experimental) undergoing neuromuscular training with K-Tape. Data collection utilizes the Numeric Pain Rating Scale (NPRS) for pain, the Star Excursion Balance Test for dynamic balance, Foot and Ankle Ability Measure (FAAM)-Sport Subscale, and a goniometer for range of motion. Participants undergo three sessions of treatment per week for four weeks. The collected data will be analyzed using SPSS version 25, aiming to provide insights into the efficacy of neuromuscular training with K-Tape as a rehabilitation strategy for ankle sprains in footballers.

DETAILED DESCRIPTION:
Ankle sprains are prevalent injuries among footballers, often leading to pain, reduced range of motion, and compromised balance. While conventional closed-chain exercises are commonly employed in rehabilitation, this study addresses the potential benefits of neuromuscular training with K-Tape. The rationale lies in the understanding that precise interventions targeting neuromuscular control may offer additional therapeutic advantages. By exploring the effects of such an intervention, this research seeks to contribute insights into optimizing rehabilitation strategies for footballers recovering from ankle sprains, aiming to enhance both short-term recovery outcomes and long-term athletic performance.

This randomized controlled trial investigates the therapeutic efficacy of neuromuscular training with K-Tape in addressing pain, range of motion (ROM), and balance in footballers with grade I and II ankle sprains. Conducted at the Pakistan Sports Board in Lahore over a six-month period from March to August 2023, the study enrolled 30 male participants aged 18-30, actively engaged in sports for a minimum of one year, with weekly training durations ranging from 15 to 20 hours. Participants were divided into two groups: Group A (Control) received closed-chain exercises, while Group B (Experimental) underwent neuromuscular training with K-Tape.

Data collection utilized comprehensive tools, including the Numeric Pain Rating Scale (NPRS) for pain assessment, the Star Excursion Balance Test for dynamic balance evaluation, the Foot and Ankle Ability Measure (FAAM)-Sport Subscale to gauge functional abilities, and a goniometer for measuring range of motion. Both groups underwent three treatment sessions per week for four weeks. Group A adhered to conventional closed-chain exercises, while Group B received the experimental intervention of neuromuscular training with K-Tape.

The collected data will undergo rigorous analysis using SPSS version 25 to discern the comparative effectiveness of closed-chain exercises and neuromuscular training with K-Tape on the specified outcome measures. The study's findings are expected to provide valuable insights into potential rehabilitation strategies for footballers with ankle sprains, contributing to the advancement of sports medicine and guiding future interventions in optimizing the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age:18-28 years
* Football Players (Playing since one year)
* Ankle Sprain Grade 1, 2
* (Squeeze Test and Talar Tilt Test) performed to diagnosis ankle sprain

Exclusion Criteria:

* Any Lower limb Musculoskeletal injury/Trauma
* Ankle or lower limb fracture (since last 6months)
* Any related systemic condition (diabetes)

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Goniometer for Range of Motion | 4 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position.
Star balance excursion test for Balance | 4 weeks
  The Star Excursion Balance Test is a reliable measure and a valid dynamic test to predict risk of lower extremity injury, to identify dynamic balance deficits in patients with lower extremity conditions, and to be responsive to training programs in healthy participants and those with lower extremity conditions.
Foot and ankle ability Measure for Functional Performance | 4 weeks
  The FAAM is a self-report measure that assesses physical function of individuals with lower leg, foot, and ankle musculoskeletal disorders. 2) Sports subscale of 8 items. For each subscale patients are asked to answer each question with a single response that most clearly describes their condition within the past week.
Numerical Rating Pain Scale for Pain | 4 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alahmari KA, Kakaraparthi VN, Reddy RS, Silvian P, Tedla JS, Rengaramanujam K, Ahmad I. Combined Effects of Strengthening and Proprioceptive Training on Stability, Balance, and Proprioception Among Subjects with Chronic Ankle Instability in Different Age Groups: Evaluation of Clinical Outcome Measures. Indian J Orthop. 2020 Jul 15;55(Suppl 1):199-208. doi: 10.1007/s43465-020-00192-6. eCollection 2021 May. PMID 34122771
- [Background] Allois R, Niglia A, Pernice A, Cuesta-Barriuso R. Fascial therapy, strength exercises and taping in soccer players with recurrent ankle sprains: A randomized controlled trial. J Bodyw Mov Ther. 2021 Jul;27:256-264. doi: 10.1016/j.jbmt.2021.03.022. Epub 2021 Apr 2. PMID 34391242
- [Background] Thompson JY, Byrne C, Williams MA, Keene DJ, Schlussel MM, Lamb SE. Prognostic factors for recovery following acute lateral ankle ligament sprain: a systematic review. BMC Musculoskelet Disord. 2017 Oct 23;18(1):421. doi: 10.1186/s12891-017-1777-9. PMID 29061135
- [Background] Faizullin I, Faizullina E. Effects of balance training on post-sprained ankle joint instability. Int J Risk Saf Med. 2015;27 Suppl 1:S99-S101. doi: 10.3233/JRS-150707. PMID 26639734
- [Background] Kim K, Jeon K. Development of an efficient rehabilitation exercise program for functional recovery in chronic ankle instability. J Phys Ther Sci. 2016 May;28(5):1443-7. doi: 10.1589/jpts.28.1443. Epub 2016 May 31. PMID 27313347
- [Background] Caldemeyer LE, Brown SM, Mulcahey MK. Neuromuscular training for the prevention of ankle sprains in female athletes: a systematic review. Phys Sportsmed. 2020 Nov;48(4):363-369. doi: 10.1080/00913847.2020.1732246. Epub 2020 Feb 28. PMID 32067546